CLINICAL TRIAL: NCT03381222
Title: Risk Factors of of Ascending Aortic Atheromatous Plaque in Thai Cardiac Surgical Patient
Brief Title: Risk Factors of Ascending Aortic Atheromatous
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaowanan Khamtuikrua, principal investigator, Mahidol University
Other Study IDs: Athe001
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Ascending Aortic Atheromatous Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: epiaoryic scan — Epiaortic scan will be performed by use L15-7i Phillips®. Ultrasound probe cover with sterile cover. Five standard epiaortic views will be collected

SUMMARY:
Background Incidence of perioperative stroke In cardiac surgery is 2.6-5.2%. Ascending aortic atheromatous plaque and stroke are strongly associated.

Propose of study To determine incidence of ascending aortic atheroma in Thai people To identify risk factors which associated with ascending aortic atheroma

Methodology After received standard general anesthesia and start sternotomy. Epiaortic scan will be performed by surgeon use L15-7i Phillips® ultrasound probe cover with sterile cover.

Five standard epiaortic views will be collected. Epiaortic clips will be review and determine about atheroma by two qualified echocardiographers. Atheroma more than third grade will defined to significant. Potential risk factors of atheroma will be gather from medical record

To assess the relationship between risk factors and atheroma a univariate analysis was performed using an unpaired t-test and a Chi-square test.

For higher accuracy regarding the impact of single risk factors, a multiple logistic regression analysis was also performed.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Schedule to cardiac surgery with sternotomy

Exclusion Criteria:

Abnormal ascending aortic anatomy such as: dissection, aneurysm

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Age ≥ 18 years and schedule to cardiac surgery with sternotomy.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of ascending aortic atheromatous plaque in Thai population | 1 year
  incidence of ascending aortic atheromatous plaque

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Siriraj hospital, Bangkok Noi, Bangkok, Thailand